CLINICAL TRIAL: NCT03221829
Title: A Retrospective Analysis of Spinal Anaesthesia for Transurethral Resection of Bladder Tumour in Elderly Patients: A Single Centre Experience From 2007 to 2017
Brief Title: A Retrospective Analysis of Spinal Anaesthesia for TURBT Procedures in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Karolina Dobrońska, MD. PhD., Medical University of Warsaw
Other Study IDs: U/2/2017
Record Dates: First submitted 2017-07-13; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Spinal Anaesthesia; Bladder Tumor; Transurethral Resection
Keywords: spinal anaesthesia; elderly patients; transurethral resection of bladder tumour
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to evaluate the safety and effectiveness of spinal anesthesia among elderly patients The basic methods for diagnosis and management of bladder cancer include endoscopic procedures (cystoscopy, trans-urethral resection of bladder tumour TURBT). The age of most patients is above 60, which increases the risk of complications during the perioperative period. Usually the leading anaesthesia method in TURBT procedures is regional, mainly spinal, anaesthesia. Although the prevalence of regional upon general anaesthesia is questioned, certain positive aspects of regional anaesthesia are indisputable. Maintaining logical communication with a patient during the procedure enables early diagnosis of complications (TUR syndrome, bladder perforation). Undeniably, regional anaesthesia ensures the best pain management in the early post-operative period. The simplicity of performing an efficacious spinal block and its cost-effectiveness are additional factors, which have contributed to the acknowledgement of the method as the standard of anaesthesia for transurethral procedures.

ELIGIBILITY:
Inclusion Criteria:

* TURBT procedure
* spinal anaesthesia
* age over 60

Exclusion Criteria:

* general anaesthesia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients that have TURBT procedure under spinal anaesthesia in the Urology Departament (Medical University of Warsaw) 2007-2017
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of spinal anaesthesia for TURBT evaluated by a number of participants that had the procedure done, without the need of conversion to general anaesthesia . | 6 months
  The investigator evaluates whether the procedure could be completely performed under spinal anesthesia

SECONDARY OUTCOMES:
The influence of the bupivacaine spinal dose on bradycardia evaluated by a heart rate measurements | 6 months
  The investigator evaluates the bupivacaine doses, heart rate and the need to give atropine
The influence of the bupivacaine dose on hypotension evaluated by the non-invasive blood pressure measurements | 6 months
  The investigator evaluates the bupivacaine doses, blood pressure and the need to give ephedrine
Experienced and non-experienced anesthetist does it influence the bupivacaine dose | 6 months
  The investigator evaluates the doses of bupivacaine spinal given by specialist, young and advanced trainee.
Experienced and non-experienced anesthetist does it influence the spinal anaesthesia success | 6 months
  The investigator evaluates the success rate of spinal anaesthesia given by specialist, young and advanced trainee.

CONTACTS AND LOCATIONS:
Locations (1):
- I Department of Anaesthesiology and Intensive Care, Medical University of Warsaw, Warsaw, Poland